CLINICAL TRIAL: NCT01869244
Title: User Experience From WOODCAST 2mm Hand Resting Splint
Brief Title: WOODCAST Hand Resting Splint - Study of User Experience
Status: Completed | Type: Observational
Sponsor: Onbone Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 152/13/03/02/2013
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hand resting splint: Patients with hand resting splint treatment

SUMMARY:
The aim of the study is to collect comments form users of new type of hand resting splint.

DETAILED DESCRIPTION:
An ecologically friendly and biodegradable wood-plastic composite cast (WOODCAST) is used as a hand resting splint in this study.

ELIGIBILITY:
Inclusion Criteria:

* patient treatment involves hand resting splint; age of patient 18 - 90 years; skills with language Finnish language (written and spoken)

Exclusion Criteria:

* decreased co-operation of the patient; patient with multiple illnesses; malignancy; an illness affecting the general health.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whos treatment involves a hand resting splint. Finnish language skills (written and spoken).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
User satisfaction | 2-4 weeks
  After using hand resting splint for two weeks, patient will fill a questionaire. In the questionaire patient is asked to assess the used splint (e.g. functional performance, visual appearance), by giving points (from 1 to 10 points). Patient will use two splints from different materials during the treatment (both of the splint will be assessed by the patient).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lindfors, PhD, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Kuntoutus Orton Oy, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information of the product — http://www.onbone.com